CLINICAL TRIAL: NCT05127148
Title: Real-world Evidence of First-line Treatment With Pediatric-like Protocol for Adolescents and Young Adults Patients Diagnosed With Philadelphia-negative Acute Lymphoblastic Leukemia
Brief Title: RWE of Pediatric-like Protocol for AYA Patients With Ph-negative ALL
Status: Recruiting | Type: Observational
Sponsor: Grupo Argentino de Tratamiento de la Leucemia Aguda (Other)
Responsible Party: Sponsor
Other Study IDs: GATLA 11-LLA Ph(-)-20 AYA
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Acute Lymphoblastic Leukemia, Adult
Keywords: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescents and young adults Ph-negative ALL patients in first-line: Adolescents and young adults patients (18-40 years old) with recent diagnosis of Ph-negative acute lymphoblastic leukemia who receive argentinian pediatric-like treatment depending on risk category.
  Interventions: Other: Evaluation of survival and toxicities in AYA Ph-negative ALL patients treating in first line depending on risk category.

INTERVENTIONS:
Other: Evaluation of survival and toxicities in AYA Ph-negative ALL patients treating in first line depending on risk category. — Evaluation of survival (event free survival and overall survival) and toxicities in AYA Ph-negative ALL patients treating in first line with argentinian pediatric-like protocol depending on risk category.

SUMMARY:
This is a multicenter, observational real world clinical trial with prospective follow up that will evaluate the treatment outcome of adolescent and young patients with ph-negative acute lymphoblastic leukemia with first-line pediatric-like protocol in Argentina.

DETAILED DESCRIPTION:
The purpose of this trial is to gather real world evidence of treatment outcomes and toxicities of AYA Ph-negative ALL patients in Argentina who receive pediatric-like treatment in first line.

The study primary endpoints are to evaluate survival (event free survival and overall survival) and toxicities of AYA Ph-negative ALL patients treating in first line with pediatric-like protocol depending on risk category.

Secondary endpoints are to evaluate survival in patients who underwent allogeneic transplantation in first remission, asparaginase toxicities, and assess central cerebrospinal fluid by flow cytometry.

Every ALL patient diagnosed in our institutions will follow our guidelines with respect to diagnosis procedures.

High-risk (HR) group was defined as presenting high risk cytogenetics/molecular findings and depending on the response achieved at different time points: bad response to prednisone at day 8, ≥ 10% blast in bone marrow on day 15, minimal residual disease (MRD) by flow cytometry ≥0.1% at day 33 and ≥0.01% at day 78 in bone marrow. No-high risk group was defined as those without any high-risk factor.

The chemotherapy regimen included pre-induction phase, induction (phase I and II), consolidation, re-intensification, central nervous system (CNS) prophylaxis and maintenance therapy or ASCT in first remission .

The initial pre-induction phase, where steroids were given for 7 days. Induction therapy, phase IA consisted of weekly vincristine and daunorubicin for 4 weeks, L-Asparaginase for 8 doses or peg-asparaginase for 2 doses and prednisone continuously for 4 weeks. Phase IB consisted cytarabine for 16 doses, cyclophosphamide for 1-2 doses and 6-mercaptopurine for 28 days.

The consolidation phase consisted of 4 doses of methotrexate and 6-mercaptopurine for 56 days for Non-High Risk patients (M phase) and two cycles of three different blocks of high dose multi chemotherapy for HR patients. Re-induction consisted in two phases similar to induction. According to risk and response to treatment, patients will be candidates to maintenance for 18 months or ASCT in first remission.

Minimal residual disease will be evaluated at least on day 33, 78, in consolidation and every thee months during maintenance treatment or previous to ASCT.

ELIGIBILITY:
Inclusion Criteria:

* Signature of the form consent for participation in the study
* Ph-negative ALL diagnosis without previous treatment.

Exclusion Criteria:

* ALL with mature B phenotype (sIg +) or with the cytogenetic alterations characteristic of ALL mature B (t (8,14), t (2, 8), t (8, 22)).
* Ph-positive ALL
* Acute leukemias of ambiguous lineage (undifferentiated or mixed phenotype).
* Patients with a history of coronary, valvular or hypertensive heart disease, that contraindicate the use of anthracyclines.
* Patients with chronic liver disease in the activity phase and / or Bilirubin> 2 mg / dl and / or transaminases 5 times the normal limit, not related to ALL.
* Patients with severe chronic respiratory failure.
* Renal failure and / or creatininemia> 2 mg / dl not related to ALL.
* Serious neurological disorders, not related to leukemic disease.
* General condition affected (grades 3 and 4), not attributable to ALL.
* Uncontrolled infection by HIV, HTLV-1, HBV, HCV.
* Patient not a candidate for treatment based on the criteria of the treating physician.
* Pregnant women will have to be evaluated by a multidisciplinary team and an ethics committee.

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: All AYA (18-40 years old) with recent diagnosis of ph-negative ALL without previous treatment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate event free survival of AYA Ph-negative ALL patients treating in first line depending on risk category. | 36 months
  Evaluate event free survival of AYA Ph-negative ALL patients treating in first line with pediatric-like protocol depending on risk category.
Evaluate overall survival of AYA Ph-negative ALL patients treating in first line depending on risk category. | 36 months
  Evaluate overall survival of AYA Ph-negative ALL patients treating in first line with pediatric-like protocol depending on risk category.
Evaluate toxicities of AYA Ph-negative ALL patients treating in first line depending on risk category. | 36 months
  Evaluate toxicities of AYA Ph-negative ALL patients treating in first line with pediatric-like protocol depending on risk category.

SECONDARY OUTCOMES:
Evaluate survival in patients who underwent allogeneic transplantation in first remission | 36 months
Evaluate asparaginase toxicities. | 36 months
Assess central cerebrospinal fluid involvement by flow cytometry. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria Moirano, Dr., Principal Investigator — Grupo Argentino de Tratamiento de la Leucemia Aguda; Isolda Fernández, Dr., Study Chair — Grupo Argentino de Tratamiento de la Leucemia Aguda; Luciana Ferrari, Dr., Principal Investigator — Grupo Argentino de Tratamiento de la Leucemia Aguda
Locations (2):
- Argentina (2):
  - Instituto Privado de Hematologia y Hemoterapia, Paraná, Entre Ríos Province
  - FUNDALEU, CABA

IPD SHARING:
Plan to Share IPD: Yes
Share study protocol
Supporting Information: Study Protocol
Time Frame: The data will become available on June 2021, and will remain available until the end of the clinical trial.